CLINICAL TRIAL: NCT06866964
Title: A Single-arm, Phase II Clinical Trial of ASPIRin to prEvent Venous Thromboembolism in Patients With Advanced Germ Cell Tumors Receiving Chemotherapy
Acronym: ASPIRE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Wake Forest Baptist (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00126906; ONC-GU-2402 (Other: Atrium Health Wake Forest Baptist Comprehensive Cancer Center); Pro00085150 (Other: Advarra IRB)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Germ Cell Tumor; Testicular Cancer
Keywords: cancer; Venous thromboembolism
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms; Neoplasms; Venous Thromboembolism | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-dose aspirin (acetylsalicylic acid [ASA]) (Experimental): ASA has been shown to reduce risk of VTE. It will be self-administered, a fixed dose of ASA (81 mg) by mouth daily for 26 weeks.
  Interventions: Drug: Low-dose ASA

INTERVENTIONS:
Drug: Low-dose ASA — 81 mg by mouth daily for 26 weeks
  Other Names: aspirin

SUMMARY:
The purpose of this study is to the 6-month Venous Thromboembolism (VTE)-free rate in participants with advanced germ cell cancer at high risk of VTE who are receiving standard of care cisplatin-based chemotherapy and low-dose acetylsalicylic acid (ASA) and compare to relevant historical controls

DETAILED DESCRIPTION:
This is a single-arm, two-stage, Phase II study designed to evaluate the 6-month VTE-free rate in participants with advanced germ cell cancer at high risk of VTE who are receiving standard of care cisplatin-based chemotherapy and low-dose ASA as compared to relevant historical controls. Stage 1 will consist of 13 participants. If at least 9 of those 13 do not experience a VTE event during the first 26 weeks on the ASA, Stage 2 will be activated. Stage 2 will enroll an additional 18 participants for a total of 31. Participants will provide their own supply of ASA. Participants will self-administer a fixed dose of ASA (81 mg) by mouth daily for 26 weeks. Participants who experience the primary endpoint of VTE will stop ASA and start standard of care anticoagulation at the direction of the treating investigator. This study will initially open as a single center study at Atrium Health Wake Forest Baptist Comprehensive Cancer Center (AHWFBCCC) and additional investigational site(s) may be added following activation at the lead site.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information
2. Age ≥ 18 years and ≤ 70 years at the time of consent
3. Histological confirmation of stage IS or IIA or higher testicular or germ cell cancer. Primary mediastinal and retroperitoneal GCT are allowed. Seminoma and non-seminoma histologies are allowed.
4. Performance Status (PS) of ECOG 0-2 at the time of enrollment
5. At least one of the following "high risk" of VTE features:

   a. Stage IIC or III or higher per AJCC 8th edition criteria i. Stage IIC - any pT/TX, N3, M0, S0-1 ii. Stage III - any pT/TX, any N, M1, SX iii. Stage IIIA - any pT/TX, any N, M1a, S0-1 iv. Stage IIIB - any pT/TX, N1-3, M0, S2 or any pT/TX, any N, M1a, S2 v. Stage IIIC - any pT/TX, N1-3, M0, S3 or any pT/TX, any N, M1a, S3 or any pT/TX, any N, M1b, any S Serum marker (S category) S criteria SX Marker studies not available or not performed S0 Marker study levels within normal limits S1 LDH < 1.5 x normal and hCG < 5000 IU/L and AFP <1000 ng/mL S2 LDH 1.5 to 10 x normal or hCG 5000 to 50,000 IU/L or AFP 1000 to 10,000 ng/mL S3 LDH >10 x normal or hCG >50,000 IU/L or AFP >10,000 ng/mL

   b. Intermediate or poor risk by IGCCCG criteria i. Intermediate risk - testis/retroperitoneal primary and no non pulmonary visceral metastases plus at least one of the following markers: AFP > 1,000 ng/mL to ≤ 10,000 ng/mL, beta-hCG > 5,000 IU/L and ≤ 50,000 IU/L, LDH >1.5 x normal and ≤ 10 x normal ii. Poor risk - mediastinal primary or non-pulmonary visceral metastases plus at least one of the following markers: AFP > 10,000 ng/mL, beta- hCG > 50,000 IU/L, LDH > 10 x normal c. Khorana score of 2 or higher i. +1 point for testicular/germ cell cancer (All patients will receive +1 for their testicular/germ cell cancer diagnosis. Thus, a patient with any other Khorana characteristic [ii-v] will meet this inclusion criteria.) ii. +1 point for platelet ≥350 x 10^9/L iii. +1 point for hemoglobin <10 g/dL iv. +1 point for leukocyte count >11 x 10^9/L v. +1 point for BMI >35 kg/m^2
6. Planning or recently started 3-4 cycles of standard of care front-line cisplatin-based chemotherapy (bleomycin, etoposide, and platinum [BEP], etoposide and cisplatin [EP], or etoposide, ifosfamide, and cisplatin [VIP]). Note: ASA should be initiated no later than 2 weeks after initiation of standard front-line chemotherapy.
7. As determined by the enrolling investigator, ability of the participant to understand and comply with study procedures for the entire length of the study
8. Ability to swallow oral medications

Exclusion Criteria:

1. Receiving chemotherapy in adjuvant setting
2. Prior VTE/PE
3. Currently taking anticoagulation or antiplatelet therapy. Non-steroidal anti-inflammatory drug (NSAID) use for pain is allowed
4. Prior indication for anticoagulation or anticoagulation contraindicated (e.g., active bleed or risk of bleeding, such as history of gastrointestinal ulcers)
5. Allergy to ASA

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism (VTE)-free | 26 weeks after initiation of standard chemotherapy
  A binary variable indicating whether the participant had zero VTE events within 26 weeks of initiation of standard chemotherapy. VTE events include objectively confirmed symptomatic or asymptomatic proximal deep-vein thrombosis in a lower limb, symptomatic deep-vein thrombosis in an upper limb or distal deep-vein thrombosis in a lower limb, symptomatic or incidental pulmonary embolism, symptomatic or incidental central catheter related thrombosis, or death from venous thromboembolism.

SECONDARY OUTCOMES:
Major Bleeding Event | 26 weeks after initiation of standard chemotherapy
  A categorical variable indicating whether the participant experienced a major bleeding event within 26 weeks of initiation of standard chemotherapy. A major bleeding event is defined by the occurrence of at least one of the following. Bleeding associated with death. Overt bleeding and associated with a decrease from baseline in hemoglobin concentration by at least 2.0 g/L or with the need for transfusion of ≥ 2 units of whole blood or red cells. Bleeding in a critical area or organ such as retroperitoneal, intracranial, intraocular, intraspinal, intraarticular or pericardial, or intramuscular with compartment syndrome as determined by the investigator.
Clinically Relevant Non-Major Bleeding | 26 weeks after initiation of standard chemotherapy
  A categorical variable indicating whether the participant experienced clinically relevant non-major bleeding within 26 weeks of initiation of standard chemotherapy. Clinically relevant non-major bleeding is defined as bleeding that leads to a medical intervention, an unscheduled contact with provider, temporary cessation of oral anticoagulants or antiplatelet agent, discomfort for the participant (such as pain) or impairment of activities of daily living.
Relapse-Free Survival (RFS) | 2 years after initiation of standard chemotherapy
  Calculated from the date of enrollment to the date of first documented evidence of recurrent disease or death, whichever occurred first. For participants who have not relapsed, RFS will be censored at the last disease status assessment. Relapse will be determined by biopsy proven recurrent non-teratoma germ cell tumor, initiation of salvage chemotherapy, or rising tumor markers unequivocally.
Overall Survival (OS) | 2 years after initiation of standard chemotherapy
  Calculated from the date of enrollment to the date of death from any cause. Participants who are alive or lost to follow up at the time of the final analysis will be censored at the last known date they were alive.

OTHER OUTCOMES:
Febrile Neutropenia Event | 26 weeks after initiation of standard chemotherapy
  A binary variable indicating whether the participant experienced a febrile neutropenia event deemed to be related to acetylsalicylic acid (ASA) treatment while receiving ASA treatment. Febrile neutropenia will be documented and graded per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Landon Brown, MD, Principal Investigator — Atrium Health Wake Forest Baptist Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Charlotte, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Aurora St. Luke's Medical Center MOB, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No